CLINICAL TRIAL: NCT02623088
Title: Long Term Effects of Positive Airway Pressure Therapies on Vascular Function in Obstructive Sleep Apnea
Brief Title: CPAP Effect on Vascular Function in Obstructive Sleep Apnea
Acronym: VNI-SOH2
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.422; 2014-A01922-45 (Other: ID RCB)
Record Dates: First submitted 2015-03-27; First posted 2015-12-07 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Endothelial dysfunction; Arterial stiffness; PAP therapies
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Bank
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAP therapies: Patients with sleep apnea syndrome treated by CPAP after respiratory and vascular assessment and followed 5-7 years, as part of a clinical research.
  Interventions: Other: PAP Therapies (CPAP)

INTERVENTIONS:
Other: PAP Therapies (CPAP) — Patients with sleep apnea syndrome treated by PAP Therapies (CPAP) after diagnosis and followed 5-7 years.
  Other Names: CPAP

SUMMARY:
Obstructive sleep apnea syndrome is responsible of endothelial dysfunction, which is a independent cardio-vascular risk factor.

Assessment of pulse wave velocity (PWV) and peripheral arterial tone (PAT) are study measurements of arterial stiffness, and are strong predictors of late cardiovascular events.

This study will compare long term evolution in arterial stiffness (PWV) and endothelial dysfunction (PAT) for patients treated by Positive Airway Pressure Therapies.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) syndrome is responsible of vascular damage. Intermittent hypoxia causes oxidative stress and low-grade inflammation. By the way of increased sympathetic outflow, it's resulting endothelial dysfunction, atherosclerosis and an increase of arterial stiffness.

Finally these mechanisms are responsible of cardiovascular comorbidities: hypertension, cardiac arrhythmias or Left ventricular dysfunction. This patients presented coronary diseases or Strokes.

OSA characterized by intermittent hypoxia, is associated with atherosclerosis and vascular inflammation. Polymorphonuclear leukocytes (PMNs) are implicated in vascular inflammation by producing oxidizing radicals and proteolytic enzymes during PMN-endothelium interactions.

Reactive oxygen species (ROS) production is increased in activated cells and after attachment, PMNs release additional ROS inducing endothelial cell injury.

Continuous positive airway pressure (CPAP) is the current "gold standard" treatment for OSA, Use of CPAP restored the respiratory flow, prevents nocturnal respiratory events and daytime symptoms.

Arterial stiffness and endothelial dysfunction are linked to obstructive sleep apnea severity with a dose-effect relationship. And meta-analyse showed significant improvements in all indices of arterial stiffness after CPAP treatment in patients with OSA.

Assessment of pulse wave velocity and peripheral arterial tone are study measurements of arterial stiffness. And are strong predictors of late cardiovascular events

The investigators will compare long term evolution in arterial stiffness (PWV) and endothelial dysfunction (Peripheral arterial tone) for patients with OSA treated by Positive Airway Pressure Therapies.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a initial visit there is 4-7 years for the VNI-SOH protocol (Réf CPP Sud-Est V: 38/2006/2)
* Male or female patient, aged 20-75 years at the initial visit there is 4 to 7 years;
* Patients with a BMI> 30kg / m2 at diagnostic;
* Patient affiliated to a social security;
* Having given its written consent to participate in the study.

Exclusion Criteria:

* Person private of liberty by judicial or administrative decision, person under legal protection measure (pregnant or nursing, patient under guardianship) Article L1121-8
* Exclusion period for further studies
* Patient died or lost sight since the initial visit there 4-7 years

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sleep apnea syndrome treated by CPAP after diagnosis and followed 5-7 years, as part of a clinical research.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Long term evolution in arterial stiffness by pulse wave velocity | 4 to 7 years from baseline assessment

SECONDARY OUTCOMES:
Endothelial dysfunction by peripheral arterial tone | 4 to 7 years from baseline assessment
Parameters of systemic inflammation : CRP us, TNF-α, IL-6 , Leptin in blood sampling | 4 to 7 years from baseline assessment
Parameters of insulin resistance : glycated hemoglobin (HbA1C), blood sugar, insulin | 4 to 7 years from baseline assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Pépin, MDPhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France